CLINICAL TRIAL: NCT03436810
Title: Effect of a Structured Progressive Task-Oriented Circuit Class Training Program With Motor Imagery on Gait Performance in Patients With Stroke: A Randomized Double Blind Balanced Parallel-Group
Brief Title: Effect of Structured Progressive Task-Oriented Circuit Class Training With Motor Imagery on Gait in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MU-CIRB 2017/178.1010
Record Dates: First submitted 2018-02-05; First posted 2018-02-19 (Actual); Results first posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Stroke; Gait, Hemiplegic
Keywords: Motor Imagery; Task-Oriented Circuit Class Training; Health Education
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic; Health Education

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will receive training programs of Motor imagery (MI) for 25 minutes and Task-Oriented Circuit Class Training (TOCCT) for 65 minutes. Overall duration of program session will be 90 minutes. Training for 3 times a week over duration of 4 weeks.
  Interventions: Procedure: Motor imagery; Procedure: Task-Oriented Circuit Class Training
- Control group (Active Comparator): The control group receives programs of Health education (HE) for 25 minutes and Task-Oriented Circuit Class Training (TOCCT) for 65 minutes. Overall duration will be 90 minutes. They will be trained for 3 times a week over duration of 4 weeks.
  Interventions: Procedure: Health education; Procedure: Task-Oriented Circuit Class Training

INTERVENTIONS:
Procedure: Motor imagery — Motor imagery (MI) will be trained for the individuals by imagination of the movement. Program of MI includes 1) body relaxation and awareness 2) visual imagery 3) kinesthetic imagery and 4) refocusing of body and environment.
  Arms: Experimental group
Procedure: Health education — Topic of Health education (HE) consists of 1) Changes caused by stroke 2) Complications after stroke 3) Emotional changes after stroke 4) Living at home after stroke 5) High blood pressure and stroke and 6) Preventing recurrent stroke.
  Arms: Control group
Procedure: Task-Oriented Circuit Class Training — Program of Task-Oriented Circuit Class Training (TOCCT) consists of warm up and perform tasks 1) Stepping forward-backward onto block 2) Stepping sideway onto block 3) Heel lifts in standing to strengthen affected planter-flexor muscles 4) Standing with a decreased base and reach for object 5) Standing up from chair, walking a short distance, and returning to chair 6) Symmetrical walking and 7) Walking at fast speed.

SUMMARY:
The objectives of the study will be General Objective is to investigate the effect of TOCCT with MI on gait performance in patients with stroke. Speific Objevtives.

Specific Objectives are to compare the effect of TOCCT with MI and TOCCT with education on the spatio-temporal and functional gait variables in patients with stroke, to investigate the spatio-temporal and functional gait variables in patients with stroke after receiving TOCCT with MI and to investigate the spatio-temporal and functional gait variables in patients with stroke after receiving TOCCT with education.

DETAILED DESCRIPTION:
This study will use a sample of convenience between the ages of 18-75 years. Forty patients with stroke from the departments of physical medicine and rehabilitation, North Okkalapa General Hospital, East General Hospital and National Rehabilitation Hospital, Yangon, Myanmar will participate in this study. The sample size was calculated using the mean value of gait speed from the previous study. Probability of type I error, apha value at 0.05 and power of 0.80 were set.

All participants will be explained about details of the study and the interventions. After that, they will be asked to sign on the written consent approving by the committee of the institution prior to participate in study. All participants will be randomly allocated the participants into the experimental (TOCCT with MI) or the control (TOCCT with health education) groups. All participants will be screened following the criteria and will be collected the demographic data.

All outcome measures will be assessed by the therapist who have been trained the outcome measures of the study. As the primary outcome measurements, spatio-temporal variables will be measured by using two dimensional motion analysis method. The protocol of this method was proved to be valid and reliability from previous pilot study. For functional gait variables, six-minute walk test will be assessed for determining walking endurance, step test will be assessed for dynamic balance, and Timed Up and Go (TUG) test will be assessed for mobility function.

As the secondary outcome measure, the strength of hip flexor, hip extensor, knee flexor, knee extensor, ankle dorsiflexor, and ankle plantarflexor muscles will be assessed by using hand-held dynamometer. Muscle spasticity will be assessed by using the Modified Ashworth Scale (MAS). The outcome measures will be assessed at the baseline, after 2 weeks and 4 weeks intervention. For the safety, the therapist will measure blood pressure, pulse rate and fatigue level in the assessments, just before the training, and rest period during the training program.

Both groups will receive the same 65 minutes structured progressive TOCCT and will receive 25 minutes of MI training for the experimental group and 25 minutes of health education for the control group. So, total training duration will be 90 minutes. Intervention program will provide 3 times a week over a period of 4 weeks.

Descriptive statistic will be used for analyze the demographic and baseline characteristics of the participants. To clarify whether the data are normally distributed, the Kolmogorov Smirnov Goodness of Fit test will be used. If data are normally distributed, two-way mixed repeated measure ANOVA will be used. If the data are not normally distributed, Friedman test will be used to compare the mean differences of the spatio-temporal measures, 6 minutes walk test, step test, TUG test, muscle strength test and muscle spasticity test. The significant level is set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* First stroke and paresis on unilateral side of the body
* Age 18 - 75 years
* Post-stroke duration 3 - 12 months
* Middle cerebral artery (MCA) involvement
* Ability to walk at least 10 meters with or without using assistance
* Functional Ambulation Category (FAC) more than or equal to 3
* Mini Mental State Examination (MMSE) more than or equal to 24
* National Institutes of Health Stroke Scale (NIHSS) lessor than 14
* MI ability by the Kinesthetic and Visual Imagery Questionnaire (KVIQ-10) more than or equal to 3

Exclusion Criteria:

* Unstable cardiopulmonary problems
* Other neurological conditions such as Parkinson's disease, Alzheimer's disease, or epilepsy
* Orthopedic and rheumatologic disorders with weight bearing pain
* Unable to communicate or unable to follow commands
* Serious cardiac conditions
* Patients with unilateral spatial neglect
* Patients with ataxic movement

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2019-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunee Bovonsunthonchai, PhD, Study Chair — Faculty of Physical Therapy, Mahidol University
Locations (1):
- University of Medical Technology, Yangon, Burma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thrift AG, Thayabaranathan T, Howard G, Howard VJ, Rothwell PM, Feigin VL, Norrving B, Donnan GA, Cadilhac DA. Global stroke statistics. Int J Stroke. 2017 Jan;12(1):13-32. doi: 10.1177/1747493016676285. Epub 2016 Oct 28. PMID 27794138
- [Background] Macko RF, Ivey FM, Forrester LW. Task-oriented aerobic exercise in chronic hemiparetic stroke: training protocols and treatment effects. Top Stroke Rehabil. 2005 Winter;12(1):45-57. doi: 10.1310/PJQN-KAN9-TTVY-HYQH. PMID 15736000
- [Background] Yang YR, Wang RY, Lin KH, Chu MY, Chan RC. Task-oriented progressive resistance strength training improves muscle strength and functional performance in individuals with stroke. Clin Rehabil. 2006 Oct;20(10):860-70. doi: 10.1177/0269215506070701. PMID 17008338
- [Background] Cicinelli P, Marconi B, Zaccagnini M, Pasqualetti P, Filippi MM, Rossini PM. Imagery-induced cortical excitability changes in stroke: a transcranial magnetic stimulation study. Cereb Cortex. 2006 Feb;16(2):247-53. doi: 10.1093/cercor/bhi103. Epub 2005 May 4. PMID 15872152
- [Background] Kim JS, Oh DW, Kim SY, Choi JD. Visual and kinesthetic locomotor imagery training integrated with auditory step rhythm for walking performance of patients with chronic stroke. Clin Rehabil. 2011 Feb;25(2):134-45. doi: 10.1177/0269215510380822. Epub 2010 Oct 13. PMID 20943715
- [Background] Balasubramanian CK, Neptune RR, Kautz SA. Variability in spatiotemporal step characteristics and its relationship to walking performance post-stroke. Gait Posture. 2009 Apr;29(3):408-14. doi: 10.1016/j.gaitpost.2008.10.061. Epub 2008 Dec 3. PMID 19056272
- [Result] Billinger SA, Arena R, Bernhardt J, Eng JJ, Franklin BA, Johnson CM, MacKay-Lyons M, Macko RF, Mead GE, Roth EJ, Shaughnessy M, Tang A; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Lifestyle and Cardiometabolic Health; Council on Epidemiology and Prevention; Council on Clinical Cardiology. Physical activity and exercise recommendations for stroke survivors: a statement for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2014 Aug;45(8):2532-53. doi: 10.1161/STR.0000000000000022. Epub 2014 May 20. PMID 24846875
- [Result] Brandstater ME, de Bruin H, Gowland C, Clark BM. Hemiplegic gait: analysis of temporal variables. Arch Phys Med Rehabil. 1983 Dec;64(12):583-7. PMID 6661021
- [Result] Jorgensen L, Crabtree NJ, Reeve J, Jacobsen BK. Ambulatory level and asymmetrical weight bearing after stroke affects bone loss in the upper and lower part of the femoral neck differently: bone adaptation after decreased mechanical loading. Bone. 2000 Nov;27(5):701-7. doi: 10.1016/s8756-3282(00)00374-4. PMID 11062359
- [Result] Verma R, Arya KN, Garg RK, Singh T. Task-oriented circuit class training program with motor imagery for gait rehabilitation in poststroke patients: a randomized controlled trial. Top Stroke Rehabil. 2011 Oct;18 Suppl 1:620-32. doi: 10.1310/tsr18s01-620. PMID 22120031
- [Result] English C, Hillier SL, Lynch EA. Circuit class therapy for improving mobility after stroke. Cochrane Database Syst Rev. 2017 Jun 2;6(6):CD007513. doi: 10.1002/14651858.CD007513.pub3. PMID 28573757
- [Result] Guillot A, Collet C. Contribution from neurophysiological and psychological methods to the study of motor imagery. Brain Res Brain Res Rev. 2005 Dec 15;50(2):387-97. doi: 10.1016/j.brainresrev.2005.09.004. Epub 2005 Nov 3. PMID 16271398
- [Result] Malouin F, Richards CL, Jackson PL, Dumas F, Doyon J. Brain activations during motor imagery of locomotor-related tasks: a PET study. Hum Brain Mapp. 2003 May;19(1):47-62. doi: 10.1002/hbm.10103. PMID 12731103
- [Result] Dunsky A, Dickstein R, Marcovitz E, Levy S, Deutsch JE. Home-based motor imagery training for gait rehabilitation of people with chronic poststroke hemiparesis. Arch Phys Med Rehabil. 2008 Aug;89(8):1580-8. doi: 10.1016/j.apmr.2007.12.039. PMID 18674992
- [Result] Zimmermann-Schlatter A, Schuster C, Puhan MA, Siekierka E, Steurer J. Efficacy of motor imagery in post-stroke rehabilitation: a systematic review. J Neuroeng Rehabil. 2008 Mar 14;5:8. doi: 10.1186/1743-0003-5-8. PMID 18341687
- [Result] Aung N, Bovonsunthonchai S, Hiengkaew V, Tretriluxana J, Rojasavastera R, Pheung-Phrarattanatrai A. Concurrent validity and intratester reliability of the video-based system for measuring gait poststroke. Physiother Res Int. 2020 Jan;25(1):e1803. doi: 10.1002/pri.1803. Epub 2019 Aug 16. PMID 31418511
- [Result] Bandinelli S, Benvenuti E, Del Lungo I, Baccini M, Benvenuti F, Di Iorio A, Ferrucci L. Measuring muscular strength of the lower limbs by hand-held dynamometer: a standard protocol. Aging (Milano). 1999 Oct;11(5):287-93. doi: 10.1007/BF03339802. PMID 10631877
- [Result] Lin PY, Yang YR, Cheng SJ, Wang RY. The relation between ankle impairments and gait velocity and symmetry in people with stroke. Arch Phys Med Rehabil. 2006 Apr;87(4):562-8. doi: 10.1016/j.apmr.2005.12.042. PMID 16571398

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The potential participants were screened according to the selection criteria of the study. The eligible participants were explained about the details of the study and the interventions. After that, the processes of taking informed consent were done.
  There was no participant who was excluded after enrollment.
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: year] | 49.90 (11.59) | 55.55 (10.74) | 52.48 (11.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 15 | 11 | 26
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 20 | 20 | 40
Region of Enrollment [Number; unit: participants]
  Myanmar | 20 | 20 | 40
Stroke characteristics [Count of Participants; unit: Participants]
  Ischemic stroke | 12 | 14 | 26
  Hemorrhage stroke | 8 | 6 | 14
  Right-sided stroke | 10 | 12 | 22
  Left-sided stroke | 10 | 8 | 18
  Mild | 12 | 14 | 26
  Moderate | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change of Gait Speed at 4 Weeks
Description: Measured by using two dimensional motion analysis
Time Frame: 4 weeks after training
Population: 40
Measure: Mean (Standard Deviation); unit: meter per second
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 20 | 20
meter per second | 0.78 (0.21) | 0.58 (0.27)

2. Primary Outcome: Change of Step Length at 4 Weeks
Description: Measured by using two dimensional motion analysis
Time Frame: 4 weeks after training
Population: 40
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 20 | 20
centimeter
  affected limb | 49.76 (6.99) | 42.07 (11.46)
  unaffected limb | 47.78 (8.37) | 41.45 (12.17)

3. Secondary Outcome: Change of Step Time at 4 Weeks
Description: measured by using two dimensional motion analysis
Time Frame: 4 weeks after training
Population: 40
Measure: Median (Inter-Quartile Range); unit: second
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 20 | 20
second
  affected limb | 0.72 [0.59 to 0.80] | 0.83 [0.62 to 0.95]
  unaffected limb | 0.53 [0.48 to 0.63] | 0.70 [0.56 to 0.84]

4. Secondary Outcome: Change of Cadence at 4 Weeks
Description: measured by using two dimensional motion analysis
Time Frame: 4 weeks after training
Population: 40
Measure: Mean (Standard Deviation); unit: steps per minute
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 20 | 20
steps per minute | 94.13 (17.09) | 78.88 (26.35)

5. Secondary Outcome: Change of 6-minute Walk Score at 4 Weeks
Description: The changed score measured by using the 6-minute walk test. The higher changed scores mean a better outcome.
Time Frame: 4 weeks after training
Population: 40
Measure: Median (Inter-Quartile Range); unit: meter
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 20 | 20
meter | 246.50 [172.50 to 335.00] | 152.50 [120.75 to 330.00]

6. Secondary Outcome: Change of Number of Step at 4 Weeks
Description: The changed score is measured by using the step test, The higher score means better outcome.
Time Frame: 4 weeks after training
Population: 40
Measure: Mean (Standard Deviation); unit: number of steps
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 20 | 20
number of steps | 12.60 (2.54) | 10.65 (2.78)

7. Secondary Outcome: Change of Timed Up and Go Score at 4 Weeks
Description: The changed score is measured by using the Timed Up and Go test. The higher of changed score mean a worse outcome.
Time Frame: 4 weeks after training
Population: 40
Measure: Median (Inter-Quartile Range); unit: second
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 20 | 20
second | 11.25 [6.63 to 15.00] | 14.01 [10.00 to 30.25]

8. Secondary Outcome: Change of Muscle Strength at 4 Weeks
Description: The change score of muscle strength is measured by the hand-held dynamometer
Time Frame: 4 weeks after training
Population: 40
Measure: Median (Inter-Quartile Range); unit: kilogram
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 20 | 20
kilogram
  hip flexor | 3.30 [3.00 to 3.78] | 2.90 [2.60 to 3.08]
  hip extensor | 3.30 [2.90 to 3.67] | 3.00 [2.80 to 3.28]
  knee flexor | 3.35 [2.40 to 3.68] | 2.70 [2.43 to 3.30]
  knee extensor | 3.75 [3.40 to 4.00] | 3.00 [2.80 to 3.30]
  ankle dorsiflexor | 2.55 [1.88 to 2.80] | 2.60 [2.20 to 3.20]
  ankle planterflexor | 2.80 [2.10 to 3.48] | 2.50 [2.08 to 2.90]

9. Secondary Outcome: Change of Muscle Tone at 4 Weeks
Description: The change score is measured by using the modified Ashworth Scale for each muscle group, the minimum and maximum scores of muscle tone are 0 and 4, respectively. A higher score of tone means a worse outcome.
Time Frame: 4 weeks after training
Population: 40
Measure: Median (Inter-Quartile Range); unit: score
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 20 | 20
score
  knee flexor | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  ankle planterflexor | 1.00 [1.00 to 2.00] | 1.00 [1.00 to 1.75]

ADVERSE EVENTS:
Time Frame: The adverse event data were collected for every participant over the 4 weeks duration of the training program.
Description: Severe adverse event means falls or incidents leading to the injury requiring hospital or general practitioner visit.
Groups:
- Control Group: The control group received programs of Health education (HE) for 25 minutes and Task-Oriented Circuit Class Training (TOCCT) for 65 minutes. Overall duration will be 90 minutes. They were trained for 3 times a week over duration of 4 weeks.
  Health education: Topic of Health education (HE) consisted of 1) Changes caused by stroke 2) Complications after stroke 3) Emotional changes after stroke 4) Living at home after stroke 5) High blood pressure and stroke and 6) Preventing recurrent stroke.
  Task-Oriented Circuit Class Training: Program of Task-Oriented Circuit Class Training (TOCCT) consisted of warm up and perform tasks 1) Stepping forward-backward onto block 2) Stepping sideway onto block 3) Heel lifts in standing to strengthen affected planter-flexor muscles 4) Standing with a decreased base and reach for object 5) Standing up from chair, walking a short distance, and returning to chair 6) Symmetrical walking and 7) Walking at fast
- Experimental Group: The experimental group received training programs of Motor imagery (MI) for 25 minutes and Task-Oriented Circuit Class Training (TOCCT) for 65 minutes. Training for 3 times a week over duration of 4 weeks.
  Motor imagery: Motor imagery (MI) was trained for the individuals by imagination of the movement. Program of MI includes 1) body relaxation and awareness 2) visual imagery 3) kinesthetic imagery and 4) refocusing of body and environment.
  Task-Oriented Circuit Class Training: Program of Task-Oriented Circuit Class Training (TOCCT) consisted of warm up and perform tasks 1) Stepping forward-backward onto block 2) Stepping sideway onto block 3) Heel lifts in standing to strengthen affected planter-flexor muscles 4) Standing with a decreased base and reach for object 5) Standing up from chair, walking a short distance, and returning to chair 6) Symmetrical walking and 7) Walking
Arm/Group | Control Group | Experimental Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/10/NCT03436810/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/10/NCT03436810/SAP_001.pdf